CLINICAL TRIAL: NCT07135622
Title: Performance of the Molecular Test Xpert MTB/RIF Ultra for Early Detection of Tuberculosis at Primary Health Care Facilities in Georgia: a Parallel Cluster Randomized Controlled Trial
Brief Title: Xpert MTB/RIF Ultra Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nestani Tukvadze (Other)
Collaborators: National Center for Tuberculosis and Lung Disease, Tbilisi, Georgia (Other)
Responsible Party: Sponsor-Investigator, Nestani Tukvadze, MD. Principal Investigator, Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: req-2019-00422
Record Dates: First submitted 2025-08-07; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Tuberculosis (TB); Pulmonary TB
Keywords: Tuberculosis; Rapid Diagnosis; Xpert/Ultra; RR/MDR-TB; COVID-19
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary; COVID-19

STUDY DESIGN:
Intervention Model Description: Pragmatic, prospective, parallel cluster randomized trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Presumptive TB cases enrolled at PHC facilities (clusters) randomized in interventional arm
  Interventions: Diagnostic Test: Xpert® MTB/RIF Ultra
- Control (Active Comparator): Presumptive TB cases enrolled at PHC facilities (clusters) randomized in the control arm
  Interventions: Other: Referral to the specialized TB clinics

INTERVENTIONS:
Diagnostic Test: Xpert® MTB/RIF Ultra — Xpert® MTB/RIF Ultra test introduced for tuberculosis diagnosis at clinical trial sites randomized to interventional arm
  Arms: Interventional
Other: Referral to the specialized TB clinics — No intervention introduced at clinical trial sites randomized to control arm, patients follow standard care: referral to specialized TB clinics
  Arms: Control

SUMMARY:
Tuberculosis (TB) is the leading cause of death caused by infectious agent globally. Estimated 10 million people get ill with TB every year and in 2022 globally there was an increase in Tuberculosis cases, first time since 2010. While in previous years, the decrease in TB numbers was reflecting the impact of disruptions to essential TB services during the COVID-19 pandemic, the increase in numbers in following years have highlighted how severe this disruptions impacted essential TB services.

Access to early diagnosis, including drug resistance testing, is essential in the cascade of care. Early diagnosis enables a timely and adequate start of treatment, reducing TB transmission and increasing the likelihood of favorable outcomes of treatment. Most of the tests that are used today to diagnose TB are slow and difficult to use. A few years ago, a new simple and sensitive test for detection of TB was introduced, the Xpert MTB/RIF. A new version of this, Xpert Ultra (Ultra) has been developed.

National Center for Tuberculosis and Lung Diseases in collaboration with Swiss Tropical and Public Health Institute is investigating whether new test Xpert / Ultra, when carried out at the Primary Health Care facilities, would help patients in getting a fast and reliable TB diagnosis in the country of Georgia.

The study will involve approximately 1600 participants. The study was approved by the local Ethics Committee of the National Center for Tuberculosis and Lung Diseases.

DETAILED DESCRIPTION:
BACKGROUND INFORMATION The use of the rapid diagnostic test Xpert MTB/RIF (Xpert) for simultaneous detection of Mycobacterium tuberculosis and Rifampicin resistance has been scaled up in recent years globally, but real-life effectiveness studies could not demonstrate the expected beneficial impact on patient important clinical outcomes such as: time to diagnosis, time to treatment initiation and mortality among others.

The ideal rapid diagnostic tool should demonstrate better sensitivity and most importantly contribute to the detection of more TB cases and decreased time to diagnosis at decentralized Health Care facilities closest to the homes of the patients.

The new highly sensitive Xpert® MTB/RIF Ultra (Ultra) assay on GeneXpert® platform have the potential to overcome the limitations of Xpert by providing molecular TB testing with an improved sensitivity operating at peripheral facilities.

The presented study will assess the clinical impact and operational characteristics of Ultra at decentralized Primary Health Care (PHC) level, compared to existing routine diagnostic algorithm based on Xpert at specialized central TB service points (TB Cabinets).

OBJECTIVES AND PURPOSE In 2010, the World Health Organization (WHO) endorsed Xpert MTB/RIF, a rapid molecular diagnostic test with good performance characteristics[2,3]. In smear-positive patients, the test has a pooled sensitivity of 89%, whereas the pooled sensitivity in smear-negative, culture-positive patients is only 67%. Specificity is excellent in both groups at 99%[4].Xpert has been successfully rolled out in most high TB burden countries. However, efficacy trials showing excellent results were not further supported by real world effectiveness studies done after implementation of test by National TB Programs. In addition, tests in most cases have not been brought to the point of care level and thus could not pose a significant change.

In 2014, the WHO convened a meeting of stakeholders to establish consensus on identifying high-priority target product profiles (TPPs) for new tuberculosis diagnostics[5]. The identified high priority TPPs included; 1) a point-of-care non-sputum-based test capable of detecting all forms of TB by identifying characteristic biomarkers or bio signatures (the biomarker test), 2) a point-of-care triage test, which should be a simple, low-cost test that can be used by first-contact health-care providers to identify those who need further testing (the triage test), 3) a point-of-care sputum-based test to replace smear microscopy for detecting pulmonary TB (the smear-replacement test) and 4) a rapid drug-susceptibility test that can be used at the microscopy-centre level of the health-care system to select first-line regimen-based therapy (the rapid DST test).

The newly developed Ultra cartridge along with GeneXpert system, both products of Cepheid, Inc. - have the potential to become the smear-replacement test as outlined in the TPPs by overcoming operational challenges and the suboptimal sensitivity of the present Xpert. The new Ultra cartridge can detect TB with sensitivity similar to standard liquid culture [6]. As shown by Dorman et al for tuberculosis case detection, sensitivity of Xpert Ultra is superior to that of Xpert in patients with paucibacillary disease and in patients with HIV. The Ultra has also enhanced ability for detection of rifampicin resistance[7]. As a downside, the higher sensitivity of Ultra leads to the detection of non-viable mycobacteria, mainly in individuals with recent history of TB. The false positive results are seen predominately in samples with small amount of bacilli ("trace call" positive) which need to be interpreted according to recommendations by the WHO and in the light of the local epidemiology[8]. Furthermore, introducing a new diagnostic technology might lead to better patient care by shorter time to diagnosis, rather than through specific improved performance characteristics[9].

The proposed project will investigate the next generation molecular test Ultra with improved sensitivity onGeneXpert platform adjusted to environmental and clinical needs at point-of-care level.

HYPOTHESES

1. Symptom-based prioritization of patients and testing with Ultra on GeneXpert platform placed at PHC facility will substantially decrease time to diagnosis and time to treatment initiation of tuberculosis patients.
2. The proportion of bacteriologically confirmed TB cases initiated on TB treatment within 7 days from study enrolment will be at least 20% higher in the intervention arm compared to control arm.
3. Ultra on GeneXpert platform performed at PHC level will decrease initial lost-to-follow up by 30%.
4. Operations characteristics of Ultra will show feasibility to be implemented at Primary Health care level.

MAIN OBJECTIVES OF THE TB DIAGNOSIS STUDY AT PHC LEVEL:

1. To assess the impact of symptom-based prioritization of patients and testing with Ultra (intervention) in comparison to the standard algorithm (control) on time to diagnosis and time to treatment initiation.
2. To determine the proportion of participants who have bacteriologically confirmed TB and have TB therapy initiated within 7 and 30 days of enrolment in intervention arm compared to the control arm.
3. To evaluate the impact of Ultra (intervention) in comparison to the standard algorithm (control) on pre-treatment loss to follow-up.
4. To investigate operational characteristics of Ultra used on GX1 and GX4 platforms in PHC facilities in Georgia.

Trial subject population

Presumptive pulmonary TB patients attending selected PHC facilities will be invited to participate in the study.

TRIAL DESIGN

1.1 Primary and secondary endpoint

Primary endpoints:

1. (i) Time from enrolment to TB diagnosis: time interval between first approach to PHC and TB diagnosis Time interval between first approach to PHC positive TB diagnosis based on laboratory results (i.e. smear, culture, Xpert, Ultra) or clinical judgement (ii) Time from enrolment to TB treatment initiation Time interval between first approach to PHC and initiation of a TB treatment
2. Proportion of participants who have bacteriologically confirmed TB and have TB therapy initiated within 7 (30) days of enrolment Numerator: Participants with positive smear, culture, Xpert or Ultra result and who are on TB treatment 7 (30)* days after enrolment Denominator: All participants of the study arm.

Secondary endpoints:

1. Number of presumptive TB cases at the PHC facility Number of people approaching PHC with cough more than two weeks.
2. Proportion of patients with early stage TB disease referred to the NCTLD TB cabinet Early stage disease will be defined as no cavitation on chest x-ray and negative smear microscopy results
3. Time from onset of symptoms to diagnosis Time interval between first TB symptom and TB diagnosis based on laboratory results (i.e. smear, culture, Xpert, Ultra) or clinical judgement

3 Proportion of patients with unfavourable outcomes after enrolment and loss to follow up measured at 6 months Unfavourable outcome is defined as lost to follow-up, death, treatment failure, and patient transfer 4 Proportion of patients with bacteriologically confirmed TB after 6 months Numerator: Participants with positive smear, culture, Xpert or Ultra result 30 days after enrolment Denominator: All participants of the study arm. 5 Proportion of patients diagnosed with TB from PHC sites Numerator: Number of all confirmed TB cases from all PHC site Denominator: Number of all confirmed TB cases diagnosed during trial period in RCT catchment area (self-referred, referred from specialized secondary, tertiary level clinics) 6 Operational characteristics of Ultra:

1. Error rates
2. Platform failure
3. User appraisal

1.2 Trial design

This is a pragmatic, prospective, parallel cluster randomized trial in PHC facilities, routine diagnostic settings of the Georgian health system.

1.3 Measure to minimize bias

The objective of the study is to assess Ultra in routine use. The study-related procedures will be embedded into the routine practice at the PHC facilities to avoid any influence by the study. Enrolment criteria will be defined identically for both intervention and non-intervention arms to avoid selection bias.

Selection of study sites will not consider factors such as urban representation. PHC facilities with rationale amount of registered beneficiaries (population attributed to receive health care at selected HCF) and number of TB suspects are located only at city levels. The capital city Tbilisi will not be considered for the study due to a different set-up of patient/sample flow in comparison to the rest of the country.

1.4 Study duration and duration of subject participation

Study duration will be 24 months:

* 1 month preparation (IRB approvals, agreement set-up)
* 3 months initiation: staff recruitment, qualitative data collection tool development, study staff training, eCRF and online database development;
* 12 months: Prospective enrolment of the patients at randomized PHC facilities; End of 12 month, collection of qualitative data on performance characteristics using specially developed data collection tool
* 6 months follow up of individual study subjects;
* 2 months data collection, analysis and distribution of study results. Manuscript publications: within three months after study completion

1.5 Recruitment

The most common symptom of Pulmonary TB "cough more than two weeks" will be a sign for "presumptive TB case". This symptom will be added to standard registration log at the entrance of every PHC facility in both intervention and control arms. Cough information along with standard registration details will be filled by registration desk.

In the intervention PHC facilities, patients with cough for more than two weeks on initial presentation will immediately be referred to the study nurse. The study nurse will obtain informed consent. All consenting patients will obtain one on spot sputum sample for further investigation with Xpert/Ultra on the site. After testing, cases with positive Ultra results will be referred to TB cabinets. Notification of positive cases will also be sent to TB cabinets and regional coordinators. In non-intervention PHC facilities, patients with "cough more than two weeks" will be added to the standard registration log at the entrance and will continue with the standard approach for examinations and referral without having Xpert Ultra testing.

All study participants from intervention and control arm will receive the same standard of care for tuberculosis diagnostics and consecutive treatment at TB cabinet level. TB diagnosis will further be confirmed with standard examinations according to National Guidelines approved by the MoH, which includes additional clinical examination, chest x-ray and laboratory examinations (culture and DST), TB treatment based on molecular or phenotypic DST and further follow up. The only difference will be: treatment will be initiated based on Ultra results in the interventional arm and on MTB/RIF results or clinical decision in control arm.

Enrolment will continue for a total of 12 months. Clinical and contact data (address, phone numbers) will be collected from participants on day 0.

1.6 Inclusion criteria

* Presumptive pulmonary TB patients, as defined by the NTP treatment guidelines.
* Adults 18 years old and above

1.7 Exclusion criteria

* Patients with symptoms which are only attributable to extra-pulmonary TB
* Patients below the age of 18 years

1.8 Criteria for discontinuation of trial site

Reasons for the early closure of a study site by investigator may include but are not limited to:

* Failure of the site staff to comply with the protocol, the requirements of the IRB/IEC or local health authorities, the sponsor's procedures, or GCP guidelines, including the failure to meet capacity requirements outlined at the start of the study.
* Inadequate recruitment of participants by the site
* Discontinuation of further study intervention development

ELIGIBILITY:
Inclusion Criteria:

* Presumptive pulmonary TB patients, as defined by the NTP treatment guidelines.
* Adults 18 years old and above

Exclusion Criteria:

* Patients with symptoms which are only attributable to extra-pulmonary TB
* Patients below the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 778 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Time from enrolment to TB diagnosis | Time interval between first approach to PHC and TB diagnosis
  Time interval between first approach to PHC and positive TB diagnosis based on laboratory results (i.e. smear, culture, Xpert, Ultra) or clinical judgement
Proportion of participants who have bacteriologically confirmed TB and have TB therapy initiated within 7 (30) days of enrolment | At 7 (30) days from bacteriological confirmation
  Numerator: Participants with positive smear, culture, Xpert or Ultra result and who are on TB treatment 7 (30) days after enrolment Denominator: All participants of the study arm.

SECONDARY OUTCOMES:
Number of presumptive TB cases at the PHC facility | At baseline
  Number of people approaching PHC with presumptive TB symptoms, ex: cough more than two weeks.
Proportion of patients with early stage TB disease | From the onset of TB symptoms till the date of diagnostic procedures (X-ray and microscopy) at specialized TB clinics
  Early stage disease defined as no cavitation on chest x-ray and negative smear microscopy results
Time from onset of symptoms to diagnosis | Time interval between first TB symptom and TB diagnosis
  Time interval between first TB symptom and TB diagnosis based on laboratory results (i.e. smear, culture, Xpert, Ultra) or clinical judgement
Proportion of patients with unfavorable outcomes | Unfavorable outcomes after enrolment and loss to follow up measured at 6 months
  Unfavorable outcome defined as lost to follow-up, death, treatment failure, and patient transfer
All-course mortality | Within 12 months from the end of last patients enrolment
  All-course mortality defined as the number of deaths from any cause within study population

CONTACTS AND LOCATIONS:
Locations (1):
- National Center for Tuberculosis and Lung Diseases, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No